CLINICAL TRIAL: NCT01467986
Title: Prospective, Open Label, Randomized Phase II Trial to Assess a Multimodal Molecular Targeted Therapy in Children, Adolescent and Young Adults With Relapsed or Refractory High-risk Neuroblastoma
Brief Title: Multimodal Molecular Targeted Therapy to Treat Relapsed or Refractory High-risk Neuroblastoma
Acronym: RIST-rNB-2011
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Selim Corbacioglu, Prof. Dr. med., University of Regensburg
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: RIST-rNB-2011
Record Dates: First submitted 2011-10-27; First posted 2011-11-09 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Neuroblastoma Recurrent
Keywords: neuroblastoma; molecular targeted therapy; protein kinase inhibitor; mTOR Inhibitor; cytostatic topoisomerase-I-inhibitor; temozolomide; irinotecan; dasatinib; rapamycin
MeSH Terms: conditions — Neuroblastoma | interventions — Dasatinib; Sirolimus; Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Irinotecan, Temozolomide (Active Comparator): Patients randomized to the control arm receive irinotecan (I) and temozolomide (T) alone.
  Interventions: Drug: Temozolomide; Drug: Irinotecan
- Rapamycin, Dasatinib, Temozolomide, Irinotecan (Experimental): Patients with rNB receive on the study arm the experimental combination of rapamycin (R)- mTOR Inhibitor, dasatinib (D)- protein kinase inhibitor irinotecan (I)- cytostatic topoisomerase-I-inhibitor and temozolomide (T)- Antineoplastic agent
  Interventions: Drug: Dasatinib; Drug: Rapamycin; Drug: Irinotecan; Drug: Temozolomide

INTERVENTIONS:
Drug: Dasatinib — Pharmacotherapeutic Group: protein kinase inhibitor ATC-Code: L01XE06 Excipients: Tablet core: Lactose monohydrate, Cellulose, microcrystalline, Croscarmellose sodium, Hydroxypropyl cellulose, Magnesium stearate. Film-coating: Hypromellose, Titanium dioxide, Macrogol 400 Formulation: film coated tablet Route of Administration: orally. Patients should be instructed to swallow the tablets as a whole and not to split, chew, or crush them.
  Other Names: Sprycel®
  Arms: Rapamycin, Dasatinib, Temozolomide, Irinotecan
Drug: Rapamycin — Pharmacotherapeutic Group: Immunosuppressive agents - mTOR Inhibitors ATC-Code: L04A A10 Excipients: Polysorbat 80, Phosal 50 PG ((3-sn-Phosphatidyl)cholin from Soy beans, Propylenglycol, lipid acid mono- and -diglyzeride from Soy oil, Ethanol (1,5% bis 2,5%), Soy liid acid and Palmitoyl ascorbic acid) Formulation: Oral solution Route of Administration:orally
  Other Names: Rapamune®
  Arms: Rapamycin, Dasatinib, Temozolomide, Irinotecan
Drug: Irinotecan — Pharmacotherapeutic Group: cytostatic topoisomerase-I-inhibitor ATC-Code: L01XX19 Excipients: Sorbitol (E420), lactic acid, sodium hydroxid (to adjust the pH to 3.5), water for injection Formulation: concentrate for solution for infusion Route of Administration: intravenously
  Other Names: Irinomedac®
  Arms: Rapamycin, Dasatinib, Temozolomide, Irinotecan
Drug: Temozolomide — Pharmacotherapeutic Group: Antineoplastic agents - Other alkylating agents, ATC-Code: L01A X03 Excipients: Capsule content: Anhydrous lactose, Sodium starch glycolate Type A, Colloida anhydrous silica, Tartaric acid, Stearic acid. Capsule shell: Gelatine, Titanium dioxide (E171).
  Printing ink: Shellac Propylene glycol, Titanium dioxide (E171), Sunset yellow FCF Aluminium Lake (E110) Formulation: capsule, hard Route of Administration: orally; Temomedac hard capsules should be administered in the fasting state. The capsules must be swallowed whole with a glass of water and must not be opened or chewed
  Other Names: Temomedac®
  Arms: Irinotecan, Temozolomide
Drug: Irinotecan — Pharmacotherapeutic Group: cytostatic topoisomerase-I-inhibitor ATC-Code: L01XX19 Excipients: Sorbitol (E420), lactic acid, sodium hydroxid (to adjust the pH to 3.5), water for injection Formulation: concentrate for solution for infusion Route of Administration: intravenously
  Other Names: Irinomedac®
  Arms: Irinotecan, Temozolomide
Drug: Temozolomide — Pharmacotherapeutic Group: Antineoplastic agents - Other alkylating agents, ATC-Code: L01A X03 Excipients: Capsule content: Anhydrous lactose, Sodium starch glycolate Type A, Colloida anhydrous silica, Tartaric acid, Stearic acid. Capsule shell: Gelatine, Titanium dioxide (E171).
  Printing ink: Shellac Propylene glycol, Titanium dioxide (E171), Sunset yellow FCF Aluminium Lake (E110) Formulation: capsule, hard Route of Administration: orally; Temomedac hard capsules should be administered in the fasting state. The capsules must be swallowed whole with a glass of water and must not be opened or chewed
  Other Names: Temomedac®
  Arms: Rapamycin, Dasatinib, Temozolomide, Irinotecan

SUMMARY:
Children, adolescents and young adults with high risk relapsed or treatment refractory neuroblastoma (rNB) represent a group of patients with dismal prognosis for whom a recommended standard salvage therapy is currently not available.

The multimodal metronomic approach combining molecular targeted drugs (rapamycin and dasatinib) with conventional chemotherapy (irinotecan and temozolomide) will be investigated in a randomized fashion as new treatment strategy for patients with rNB. The intention is to assess the therapeutic benefit of molecular targeted drugs for the treatment of rNB.

The combination of irinotecan and temozolomide showed activity in the treatment of several solid organ tumors, brain tumors and neuroblastoma. In one study rNB patients received a median of 5 courses of 5 days irinotecan and temozolomide every 3 to 4 weeks with a cumulative dose of 35% lower than in the RIST design. 33% had disease regression with 8% CR or PR. A phase II study in rNB also using irinotecan and temozolomide with a substantially lower intensity showed a response rate of 15%.

The combination of a mTOR inhibitor with a multi-kinase inhibitor demonstrated in preclinical studies a synergistic effect on cell cycle arrest, apoptosis and sensitization for radio- and chemotherapy. It is assumed that this combination of molecular targeted drugs with a tolerable conventional chemotherapy consisting of irinotecan and temozolomide can substantially improve the outcome of this patient population. A group of 20 rNB patients treated with the RIST therapy approach in a compassionate use setting showed an overall survival of 55% at a median of 80 weeks with a tolerable adverse event profile.

ELIGIBILITY:
Inclusion Criteria:Patients with relapsed high-risk neuroblastoma (stage IV and all MYCN pos. stages) or progressive disease during primary treatment (=rNB) and all of the following criteria will be considered for admission to the clinical trial:

* Children, adolescents and young adults less than 25 years
* Signed written informed consent
* Females of childbearing age must have a negative urine pregnancy test prior to starting the study drug. The first pregnancy test must be performed within 10-14 days prior to the start of the study drug and the second pregnancy test must be performed within 24 hours prior to the start of study drug. The subject may not receive the study drug until the investigator has verified that the results of these pregnancy tests are negative.
* Females of childbearing age must comply with the institutional standards of birth control with a pearl index <1%. Contraception must be started at least four weeks before the start of the investigational therapy.
* Females of childbearing age must be willing to abstain from breastfeeding for the duration of the clinical trial and for at least 30 days after discontinuation of the clinical trial.
* Males must agree not to father a child and must use latex condom during any sexual contact with women of childbearing age during and for 6 months after therapy ends or is stopped, even if they have undergone successful vasectomy.
* Willing and able to complete the clinical trial procedures, as described in the protocol
* Non-smoker for at least the previous 3 months. Smoking is not allowed during the entire study period
* Abstain from alcohol within the last 24 hours before screening and before admission to the clinical trial center as well as during the entire clinical trial. The regular daily ethanol intake has to be less than 20g/day for at least the previous three month.
* Patients are required to have an absolute neutrophil count (ANC) ≥ 500/µL, hemoglobin ≥8g/dL (transfusion permitted), and an unsupported platelet count ≥30,000/µL unless:

  1. extensive bone marrow involvement was documented
  2. patient is refractory or relapsed early after primary therapy

Exclusion Criteria:

* Pregnancy, nursing
* Patients who suffered from a thrombotic event and need anticoagulation (i.e. coumadin derivatives or low molecular weight heparin derivatives, LMWH)
* Patients with cardiac arrhythmias especially prolonged QT
* Patients with chronic inflammatory bowel diseases and/or bowel obstruction
* Patients with bilirubin serum levels 1,5 fold above the upper normal limit
* Vaccination with a live virus vaccine during the clinical trial
* Impaired liver function and/or impaired renal function (hepatic and renal index parameter two times above normal range; see below)
* Potentially unreliable subjects, probably non compliant subjects and those judged by the investigator to be unsuitable for the study
* Doubts about the patient's cooperation
* Any contraindications or known hypersensitivity to the IMPs or to any of the other components: (see SPC ("Fachinformation", appendix)
* Known allergic reactions to the treatment medication
* Patients who were treated with radiation and/or chemotherapy for any other oncological condition
* Participation in any other phase I to III trial
* Sexually active patients who refuse to use contraception according to the institutional requirements
* Patients with extremely poor general condition (Karnofsky or Lansky score <50%)
* Neutrophil count (ANC) <500/µL, hemoglobin <8g/dL (transfusion permitted), and an unsupported platelet count <30 000/µL
* 12-lead ECG with QTc>500 msec / QTc>60 msec baseline
* Patients with hepatitis B reactivation

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2013-08; Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is progression-free survival (PFS) | Time interval from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 52 weeks
  The primary objective of this trial is the evaluation of progression-free survival of rNB in children, adolescents and young adults, comparing a multimodal treatment regimen consisting of temozolomide (T), irinotecan (I), rapamycin (R) and dasatinib (S) against irinotecan (I) and temozolomide (T) (I/T) alone

SECONDARY OUTCOMES:
Overall survival (OS) | Response to the investigational treatment after 4 courses and 8 courses of I/T and 1-year-follow-up
Response to the investigational treatment after 4 and 8 courses of I/T and 1-year-follow-up in the RIST treatment arm | Response to the investigational treatment after 4 courses and 8 courses of I/T and 1-year-follow-up
Duration until adequate response to this treatment regimen | Response to the investigational treatment after 4 courses and 8 courses of I/T and 1-year-follow-up
Assessment of quality of life (Lansky and Karnofsky Scores) | • Response to the investigational treatment after 4 courses and 8 courses of I/T and 1-year-follow-up
Toxicity of this combination of drugs in children, adolescents and young adults with rNB | From the first course of the investigational treatment up to the end of the trial assessed to 52 weeks.
  Assessment according to the latest version of the CTC criteria. In particular due to the expected AE Profile:
  * Myelosuppressive measures (RBC, PLT units)
  * Infectious complications
  * Gastrointestinal problems
Safety and tolerability of the investigational treatment | Response to the investigational treatment after 4 courses and 8 courses of I/T and 1-year-follow-up
  Assessment according to the latest version of the CTC criteria. In particular due to the expected AE Profile:
  * Myelosuppressive measures (RBC, PLT units)
  * Infectious complications
  * Gastrointestinal problems
Assessment of the prognostic relevance of International Neuroblastoma Risk Group (INRG) classification system on the event free survival | Response to the investigational treatment after 4 courses and 8 courses of I/T and 1-year-follow-up
Prognostic relevance of defined factors on the event free survival in this patient population (i.e. response assessment of HVA, VMA, NSE) | Response to the investigational treatment after 4 courses and 8 courses of I/T and 1-year-follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Selim Corbacioglu, MD, Principal Investigator — University of Regensburg, Department of Pediatric Hematology and Oncology
Locations (1):
- University Hospital Regensburg, Department of Pediatric Hematology and Oncology, Regensburg, Germany

REFERENCES:
- [Derived] Corbacioglu S, Lode H, Ellinger S, Zeman F, Suttorp M, Escherich G, Bochennek K, Gruhn B, Lang P, Rohde M, Debatin KM, Steinbach D, Beilken A, Ladenstein R, Spachtholz R, Heiss P, Hellwig D, Troger A, Koller M, Menhart K, Riemenschneider MJ, Zoubaa S, Kietz S, Jakob M, Sommer G, Heise T, Hundsdorfer P, Kuhnle I, Dilloo D, Schonberger S, Schwabe G, von Luettichau I, Graf N, Schlegel PG, Fruhwald M, Jorch N, Paulussen M, Schneider DT, Metzler M, Leipold A, Nathrath M, Imschweiler T, Christiansen H, Schmid I, Crazzolara R, Niktoreh N, Cario G, Faber J, Demmert M, Babor F, Frohlich B, Bielack S, Bernig T, Greil J, Eggert A, Simon T, Foell J. Irinotecan and temozolomide in combination with dasatinib and rapamycin versus irinotecan and temozolomide for patients with relapsed or refractory neuroblastoma (RIST-rNB-2011): a multicentre, open-label, randomised, controlled, phase 2 trial. Lancet Oncol. 2024 Jul;25(7):922-932. doi: 10.1016/S1470-2045(24)00202-X. PMID 38936379